CLINICAL TRIAL: NCT01977625
Title: Utilizing fMRI to Determine the Effects of Vyvanse® on Memory, Attention, and Brain Activity in Menopausal Women
Brief Title: LDX and Functional Magnetic Resonance Imaging (fMRI in Menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 814735
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2017-07

CONDITIONS: Menopause; Brain Activity; Cognition
Keywords: Menopause; fMRI; Vyvanse
MeSH Terms: interventions — Lisdexamfetamine Dimesylate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine (Active Comparator): Lisdexamfetamine or Vyvanse
  Interventions: Drug: Lisdexamfetamine
- Sugar Pill (Placebo Comparator): Placebo pill, capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine — The overall objective of this study is to assess the effects of LDX on brain activation patterns during tasks of sustained attention and working memory in menopausal women.
  Other Names: Vyvanse®
  Arms: Lisdexamfetamine
Other: Placebo — To assess the effects of a placebo pill on brain activation patterns during tasks of sustained attention and working memory in menopausal women.
  Other Names: Sugar pill
  Arms: Sugar Pill

SUMMARY:
This study seeks to assess the effects of lisdexamfetamine (trademark name: Vyvanse; LDX) on executive function and prefrontal cortex activation in menopausal women ages 45-57, who report subjective cognitive difficulties. This protocol will recruit women from Dr. Epperson's ongoing study, Protocol #812470, to examine the impact of LDX on brain activation during performance of cognitive tasks specifically probing prefrontal cortex function.

ELIGIBILITY:
Inclusion Criteria:

1. Have no previous or present history of a DSM-IV psychiatric or substance dependence disorder within the previous year, according to the Structured Clinical Interview for Diagnosis- DSM-IV (SCID)-Non-Patient Version;
2. Are within 5 years of last menstrual period (LMP);
3. Have a follicular stimulating hormone level (FSH) of 20 IU/ml;
4. Are able to give written informed consent;
5. Must have clear urine toxicology screen upon recruitment;
6. Are fluent in written and spoken English;
7. Are right-handed;
8. Negative urine pregnancy test if still menstruating.

Exclusion Criteria:

1. Mini-mental status exam score of less than or equal to 24;
2. Presence of a psychiatric disorder within previous year or a life time history of ADHD or psychotic disorder including bipolar disorder, schizoaffective disorder, and schizophrenia;
3. Lifetime history of drug addiction or abuse, except nicotine;
4. Regular use of other psychotropic medication;
5. Regular use (more than once a week) of alcohol that is less than 3 drinks/day;
6. Presence of a contraindication to treatment with stimulant medication unless the condition is controlled with medication; this would include the presence of uncontrolled hypertension, coronary disease, atrial fibrillation, and arrhythmia;
7. History of seizures;
8. History of cardiac disease including known cardiac defect or conduction abnormality;
9. Abnormal electrocardiogram during screening;
10. Use of estrogen therapy within previous 2 months;
11. Current pregnancy or planning to become pregnant;
12. Metallic implant;
13. Claustrophobia.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Neill Epperson, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Penn Center for Womens Behavioral Wellness, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epperson CN, Pittman B, Czarkowski KA, Bradley J, Quinlan DM, Brown TE. Impact of atomoxetine on subjective attention and memory difficulties in perimenopausal and postmenopausal women. Menopause. 2011 May;18(5):542-8. doi: 10.1097/gme.0b013e3181fcafd6. PMID 21293309
- [Result] Epperson CN, Shanmugan S, Kim DR, Mathews S, Czarkowski KA, Bradley J, Appleby DH, Iannelli C, Sammel MD, Brown TE. New onset executive function difficulties at menopause: a possible role for lisdexamfetamine. Psychopharmacology (Berl). 2015 Aug;232(16):3091-100. doi: 10.1007/s00213-015-3953-7. Epub 2015 Jun 11. PMID 26063677
- [Result] Shanmugan S, Loughead J, Nanga RP, Elliott M, Hariharan H, Appleby D, Kim D, Ruparel K, Reddy R, Brown TE, Epperson CN. Lisdexamfetamine Effects on Executive Activation and Neurochemistry in Menopausal Women with Executive Function Difficulties. Neuropsychopharmacology. 2017 Jan;42(2):437-445. doi: 10.1038/npp.2016.162. Epub 2016 Aug 23. PMID 27550732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 participants were recruited from the parent study NCT01324024 to complete 3 brain imaging scans.
Pre-assignment Details: Of the 18 participants who were recruited, they all were deemed eligible based on the criteria for the parent study NCT01324024. In addition, they must have been deemed eligible to undergo a functional brain imaging scan. Of these 18 participants, 14 completed all 3 scans.
Groups:
- Lisdexamfetamine, Then Placebo: Participants first received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks followed by a 2-week washout, then they received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks.
- Placebo, Then Lisdexamfetamine: Participants first received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks followed by a 2-week washout, then they received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks..
Period: First Intervention (4 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo, Then Lisdexamfetamine
Started | 11 | 7
Completed | 8 | 7
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0
Period: Washout (2 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo, Then Lisdexamfetamine
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo, Then Lisdexamfetamine
Started | 8 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of the 18 participants who were recruited, they all were deemed eligible based on the criteria for the parent study NCT01324024. In addition, they must have been deemed eligible to undergo a functional brain imaging scan. Analysis of the participants presented below is indicative of the 14 participants who successfully completed all 3 scans.
Groups:
- All Participants: Participants first received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks followed by a 2-week washout, then they received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [49 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Blood Oxygen Level Dependent (BOLD) Signal
Description: Blood-oxygen-level dependent contrast imaging, or BOLD-contrast imaging, is a method used in functional magnetic resonance imaging (fMRI) to observe different areas of the brain or other organs, which are found to be active at any given time. BOLD signals were compared from baseline, first intervention and second intervention.
Time Frame: 10 weeks
Population: All participants who completed all phases of the study were included in the outcome analysis.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo: Placebo pill, capsules
  Placebo: To assess the effects of a placebo pill on brain activation patterns during tasks of sustained attention and working memory in menopausal women.
Arm/Group | Lisdexamfetamine | Placebo
Number analyzed (Participants) | 14 | 14
percent change | 0.41 (0.65) | -0.11 (0.46)

2. Secondary Outcome: Change in BADDS Total Score
Description: The total BADDS ranged from 0-120 with higher scores meaning greater problems with memory, attention and focus. Difference in BADDS score from Baseline to End of Treatment for each study Arm was calculated.
Time Frame: 10 weeks
Population: Participants who completed all 3 scans.
Measure: Mean (Standard Deviation); unit: change in units
Groups:
- Lisdexamfetamine; Placebo: 14 participants completed all 3 scans.
Arm/Group | Lisdexamfetamine | Placebo
Number analyzed (Participants) | 14 | 14
change in units | -23.36 (11.57) | -8.57 (12.51)

ADVERSE EVENTS:
Groups:
- Lisdexamfetamine: Participants first received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks followed by a 2-week washout, then they received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks.
- Placebo: Participants first received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks followed by a 2-week washout, then they received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks.
Arm/Group | Lisdexamfetamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine (N=15) | Placebo (N=15)
Increase heart rate (Cardiac disorders) | 1 (1) | 0 (0)
Increase blood pressure (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes